CLINICAL TRIAL: NCT04232826
Title: A Clinical Trial of CNCT19 Cells in the Treatment of CD19 Positive Relapsed or Refractory Diffuse Non-Hodgkin Lymphoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Juventas Cell Therapy Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HY-CD19 CART-002
Record Dates: First submitted 2020-01-11; First posted 2020-01-18 (Actual); Last update posted 2023-03-28 (Actual); Status verified 2023-03

CONDITIONS: Diffuse Non-Hodgkin Lymphoma

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single dose of CNCT19 (Experimental): A conditioning chemotherapy regimen of fludarabine and cyclophosphamide will be administered followed by investigational treatment, CNCT19.
  Interventions: Biological: single dose of CNCT19

INTERVENTIONS:
Biological: single dose of CNCT19 — Dose A: 1.00 x 10^8 autologous CNCT19 transduced cells via intravenous infusion. Drug: Fludarabine Drug: Cyclophosphamide
  Dose B: 2.00 x 10^8 autologous CNCT19 transduced cells via intravenous infusion. Drug: Fludarabine Drug: Cyclophosphamide
  Dose C: 4.00 x 10^8 autologous CNCT19 transduced cells via intravenous infusion. Drug: Fludarabine Drug: Cyclophosphamide

SUMMARY:
This is a single arm, open-label, non-randomized, dose-escalation, phase I study to determine the safety and efficacy of CNCT19 in adult patients with relapsed or refractory diffuse Non-Hodgkin lymphoma.

DETAILED DESCRIPTION:
This is a single arm, open-label, non-randomized, dose-escalation, phase I study to determine the safety and efficacy of CNCT19 in adult patients with relapsed or refractory diffuse Non-Hodgkin lymphoma. The study will have the following sequential phases: Screening, Pre-Treatment (Cell Product Preparation & Lymphodepleting Chemotherapy), Treatment and Follow-up, and Survival Follow-up. The total duration of the study is 2 years from CNCT19 cell infusion.

ELIGIBILITY:
Inclusion criteria:

1. Informed consent is signed by the subject.
2. Age 18 to 75.
3. Relapsed or refractory NHL with CD19-positive after at least two systemic lines of therapy

   a. Diffuse large B cell lymphoma (DLBCL) non-specific (NOS), T-cell / Histiocyte Rich large B-cell lymphoma, elderly EBV-positive diffuse large B-cell lymphoma, primary mediastinal large B-cell lymphoma (PMBCL), chronic inflammation-associated DLBCL, follicular lymphoma (FL) transformed large B-cell lymphoma, high-grade B-cell lymphoma with MYC and BCL2 and / or BCL6 rearrangement and High-grade B-cell lymphoma-unspecified; b. Chemotherapy-refractory disease, defined as one of more of the following:
   * No response to last line of therapy; i. Progressive disease (PD) as best response to most recent therapy regimen; ii. Stable disease (SD) as best response to at least 4 courses of first-line treatment / at least 2 courses of end-line treatment (2 lines and above) with duration no longer than 6 month from last dose of therapy OR;
   * Refractory post-autologous stem cell transplant (ASCT); i. Disease progression or relapsed less than or equal to 12 months of ASCT (must have biopsy proven recurrence in relapsed individuals); ii. If salvage therapy is given post-ASCT, the individual must have had no response to or relapsed after the last line of therapy; Any BM relapse after autologous stem cell transplantation (ASCT); c. Individuals must have received two systemic lines of therapy
   * anti-CD20 monoclonal antibody unless investigator determines that tumor is CD20-negative;
   * an anthracycline containing chemotherapy regimen;
   * FL-transformed DLBCL must have received pre-chemotherapy for FL and become resistant after conversion to DLBCL.
4. At least one measurable lesion, defined as at least 1 lymph node >1.5 cm in the longest diameter, per revised IWG Response Criteria.
5. Any previous systemic immune checkpoint therapy (such as anti-PD1 / PD-L1 monoclonal antibody, etc.), at least 3 half-lives away from the Cell Product Preparation; other systemic treatments should be stoped at least 2 weeks or 5 half-lives before Cell Product Preparation (shorter Whichever comes first).
6. Eastern cooperative oncology group (ECOG) performance status of 0 to 1.
7. Sufficient bone marrow reserves defined as:

   1. Absolute neutrophil (ANC) > 1,000 / mm3;
   2. Lymphocyte absolute value (ALC) ≥ 100 / mm3;
   3. Platelet (PLT) ≥ 50,000 / mm3.
8. Adequate organ function defined as:

   1. aspartate aminotransferase (AST) ≤ 3 upper limit of normal (ULN);
   2. Serum alanine aminotransferase (ALT) ≤ 3 upper limit of normal (ULN);
   3. Total bilirubin ≤ 2 ULN, except in individuals with Gilbert's syndrome; Note: Patients with Gilbert's syndrome that bilirubin ≤ 3 ULN and direct bilirubin ≤ 1.5 ULN will be eligible;
   4. A serum creatinine≤ 1.5 ULN or Creatine removal rate ≥ 60mL/min (Cockcroft and Gault);
   5. Must have a minimum level of pulmonary reserve as ≤ Grade 1 dyspnea and oxygen saturation > 91% on room air;
   6. International normalized ratio (INR) ≤ 1.5 ULN and activated partial thromboplastin time (APTT) ≤ 1.5 ULN;
9. Non-hematological toxic reactions (excluding diseases related) caused by previous treatment were restored to ≤ 1 level before screening (excluding ≤ 2 level of neurotoxicity caused by hair loss and chemotherapy drugs).
10. Women of childbearing age have a negative blood / urine pregnancy test within 7 days before the CNCT19 infusion. Women of child-bearing potential and all male participants must use highly effective methods of contraception throughout the study and for a period of at least six months after the CNCT19 infusion.

Exclusion criteria:

1. Active CNS involvement by malignancy.
2. Patients who received chemotherapy within 2 weeks before CNCT19 infusion. The following situations are excluded:

   1. Lymphodepleting Chemotherapy prescribed by the protocol;
   2. CNS prophylaxis treatment must be stopped > 1 week prior to CNCT19 infusion.
3. Has had treatment with any prior anti-CD19 therapy.
4. Plans to receive autologous stem cell transplantation (ASCT) within 6 weeks before the CNCT19 infusion.
5. Patients who have previously received Allogeneic Hematopoietic Stem Cell Transplantation (allo-HSCT).
6. Patients with systemic vasculitis (such as Wegener granulomatosis, nodular polyarteritis, systemic lupus erythematosus) and active or uncontrolled autoimmune disease (such as autoimmune hemolytic anemia, etc.).
7. Patients who are positive for any of HBsAg, HCV-Ab, TP-Ab.
8. Patients who have previously received surgery within 4 weeks before the screening that was unsuitable for enrollment by the investigator's assessment.
9. Prior malignancy, except carcinoma in situ of the skin or cervix treated with curative intent and with no evidence of active disease. Patients with Prior malignancy that has been cured for ≥ 2 years are excluded.
10. a. Left Ventricular Ejection Fraction (LVEF) ≤45%; b. III/IV congestive heart failure (NYHA); c. Severe arrhythmia (except for Atrial fibrillation, Paroxysmal supraventricular tachycardia); d. QTc≥450ms (male)or QTc≥470ms (female)(QTcB=QT/RR1/2); e. Myocardial infarction or Coronary Artery Bypass Graft Surgery, heart stent surgery < 6 months prior to CNCT19 infusion; f. Clinically significant valvular disease; g. Other heart diseases that have been judged by the investigator to be unsuitable for receiving cell therapy.
11. Clinically significant pleural effusion.
12. Patients with a history of epilepsy, cerebrovascular ischemia / hemorrhage, cerebellar disease or other active central nervous system diseases.
13. Lymphoma affects the atrium or ventricle.
14. Clinical emergencies (such as intestinal obstruction or vascular compression) that requires urgent treatment due to obstruction or compression of lymphoma tumors during screening.
15. History of deep vein thrombosis or pulmonary embolism within 6 months of screening.
16. Known history of hypersensitivity to ingredients used in the drug.
17. Has had treat with live vaccine within 6 weeks prior to screening.
18. Patients with evidence of currently uncontrollable serious active infections (e.g., sepsis, bacteremia, fungemia, viremia, etc.).
19. Life expectancy < 12 weeks.
20. Patient in other interventional clinical studies within 3 months before the CNCT19 infusion, who have received active drug therapy, or who intend to participate in another clinical trial or receive anti-tumor therapy outside the protocol during the entire study.
21. Patients with other conditions making the patients unsuitable for receiving cell therapy as judged by the investigator.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2020-01-15 (Actual); Primary Completion 2021-01-01 (Actual); Study Completion 2022-11-01 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD), Dose Limiting Toxicity (DLT) and Recommended Phase II Dose (RP2D) | 28 days
  Determine the MTD and DLT of CNCT19 in the Treatment and recommend the dose for Phase II study.
Safety of CNCT19 therapy: CTCAE v5.0 | 24 months
  Safety measures include adverse events as assessed by CTCAE v5.0.

SECONDARY OUTCOMES:
Overall Remission Rate (ORR), which includes Complete Remission (CR) and Partial Remission (PR) | 3 months
  Efficacy of CNCT19 as measured by ORR during the 3 months after CNCT19 infusion, which includes CR and PR.
Overall Remission Rate (ORR), which includes Complete Remission (CR) and Partial Remission (PR) | 28 days
  Efficacy of CNCT19 as measured by ORR during the 28 days after CNCT19 infusion, which includes CR and PR.
Overall Remission Rate (ORR), which includes Complete Remission (CR) and Partial Remission (PR) | 2 months
  Efficacy of CNCT19 as measured by ORR during the 2 months after CNCT19 infusion, which includes CR and PR.
Overall Remission Rate (ORR), which includes Complete Remission (CR) and Partial Remission (PR) | 6 months
  Efficacy of CNCT19 as measured by ORR during the 6 months after CNCT19 infusion, which includes CR and PR.
Best Overall Response (BOR) | 24 months
  The best overall response after CNCT19 infusion.
Time to initial Response (TTR) | 6 months
  TTR is defined as the time from the CNCT19 infusion to the first documented CR or PR.
Progression-free survival (RFS) | 24 months
  PFS is defined as the time from the signing of informed consent form to the date of the documented progressive disease(PD) or death due to any cause.
Duration of remission (DOR) | 24 months
  DOR is defined as the time from the first documented CR or PR to the date of the first documented relapse or PD.
Overall survival (OS) | 24 months
  OS is defined as the time from the signing of informed consent form to the date of the last survival follow-up or death due to any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Dehui Zou, Dr., Principal Investigator — Institute of Hematology & Blood Diseases Hospital, China
Locations (2):
- China (2):
  - Henan Cancer Hospital, Zhengzhou, Henan
  - Institute of Hematology & Blood Diseases Hospital, Tianjin